CLINICAL TRIAL: NCT03811119
Title: MANTA™ Versus Suture-based Closure After Transcatheter Aortic Valve Implantation Trial
Acronym: MASH-TAVI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Nicolas van Mieghem, Principal Investigator, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MASH TAVI 06-09-2018
Record Dates: First submitted 2019-01-17; First posted 2019-01-22 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Aortic Valve Stenosis
Keywords: Vascular Closure Devices; Transcatheter Aortic Valve Implantation
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Intervention Model Description: Open label randomized trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- MANTA vascular closure device (Active Comparator): Arteriotomy closure with a collagen-based vascular closure device (MANTA™)
  Interventions: Device: MANTA vascular closure device
- Suture based vascular closure device (Active Comparator): Arteriotomy closure with 2 or more suture-based vascular closure devices (ProGlide)
  Interventions: Device: Suture based vascular closure device

INTERVENTIONS:
Device: MANTA vascular closure device — Collagen based vascular closure device
  Arms: MANTA vascular closure device
Device: Suture based vascular closure device — Suture based vascular closure device (ProGlide)
  Arms: Suture based vascular closure device

SUMMARY:
To investigate whether the collagen-based MANTA vascular closure device (VCD) is superior to suture-based VCDs in preventing vascular access site complications in patients undergoing transfemoral transcatheter aortic valve replacement.

DETAILED DESCRIPTION:
see summary

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective transfemoral TAVI for severe aortic valve stenosis with any commercially-available transcatheter heart valve (THV)
* Common femoral artery diameter > 5.0mm (14 - 22F compatible)

Exclusion Criteria:

* Symptomatic leg ischaemia
* Previous thromboendarterectomy or plastic patch of the common femoral artery
* Previous implantation of a suture-based VCD less than 30 days before, or a plug-based VCD within 6 months
* Unilateral or bilateral lower extremity amputation
* Systemic infection or a local infection at or near the access site
* Allergy to the components any of both devices (i.e. bovine materials or any other device material, including collagen and/or collagen products, polyglycolic or polylactic acid, stainless steel or nickel)
* Active bleeding or bleeding diathesis including thrombocytopenia (platelet count <50,000 cells/UL), thrombasthenia, hemophilia, or von Willebrand disease
* Patients in whom continuous oral anticoagulation therapy cannot be stopped for the peri-procedural period or patients with INR >1.8 at the time of the procedure
* Patient unable to be adequately anti-coagulated for the procedure
* Morbidly obese or cachectic (BMI >40 kg/m2 or <20 kg/m2)
* Anatomical and procedural contraindication for suture-based or Manta closure (lack of proper puncture site in the common femoral artery in terms of calcification, size, and atherosclerotic disease)
* Absence of computed tomographic data of the access site before the procedure
* Patient cannot adhere to or complete the investigational protocol for any reason including but not limited to geographical residence, psychiatric condition or life threatening disease
* Known pregnancy at time of randomization (in women of childbearing potential a negative pregnancy test is mandatory)
* Participating in trials in which the primary endpoint includes bleeding or vascular complications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2018-10-30 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Composite rate of major- and minor vascular complications according to VARC-2 | Between transcatheter aortic valve implantation and 30 days follow-up
  The primary endpoint will consist of the composite of major- and minor vascular complications according to the Valve Academic Research Consortium (VARC)-2 at 30 days follow-up.

SECONDARY OUTCOMES:
Number of Participants with a Major Vascular Complication according to VARC-2 | Between transcatheter aortic valve implantation and 30 days follow-up
  total number of participants major vascular complications
Number of Participants with a Minor Vascular Complication according to VARC-2 | Between transcatheter aortic valve implantation and 30 days follow-up
  total number of participants minor vascular complications
All-cause death rate | Between transcatheter aortic valve implantation and 30 days follow-up
  A distinction between cardiac-, non-cardiac vascular and non-cardiovascular death will be made
Number of Participants with a major- or life threatening bleeding according to VARC-2 | Between transcatheter aortic valve implantation and 30 days follow-up
  total number of participants with major/life-threatening bleedings
Need for transfusions for access site related bleeding/complications | Between transcatheter aortic valve implantation and 30 days follow-up
  Total number of transfusions of RBC because of site-related bleeding
Number of Participants with vascular closure device failure | Between transcatheter aortic valve implantation and 30 days follow-up
  Failure of a closure device to achieve haemostasis at the arteriotomy site leading to alternative treatment (other than manual compression or adjunctive endovascular ballooning)
Time to hemostasis | During the TAVI procedure
  After the use of a vascular closure device the time to hemostasis will be classified as immediate hemostasis, hemostasis after 5 minutes manual compression, hemostasis after 10 minutes manual compression, hemostasis after endovascular ballooning, hemostasis after endovascular intervention or hemostasis after surgical intervention
Total procedure time | During the TAVI procedure
  The total procedural time in minutes will be compared between the two treatment arms
Number of Participants with a clinically relevant bleeding defined as BARC 2, 3 and 5 | Between transcatheter aortic valve implantation and 30 days follow-up
  Clinically relevant bleeding defined as BARC 2, 3 and 5
Length of hospital stay | Up to a maximum of 30 days after the TAVI procedure
  The total length of hospital stay in days will be compared between the two treatment arms

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas M Van Mieghem, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus University Medical Center Rotterdam, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No
no sharing of individual data (no permission from participants. GDPR)